CLINICAL TRIAL: NCT02388659
Title: Clinical Development of Cancer-Specific MRS Biomarkers in Malignant Gliomas
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: STU022014-048; R01CA184584 (NIH)
Record Dates: First submitted 2015-02-19; First posted 2015-03-17 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Malignant Gliomas; Oligodendrogliomas; Astrocytomas
Keywords: MRS Biomarkers
MeSH Terms: conditions — Glioma; Oligodendroglioma; Astrocytoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain MRI/MRS Patients: 3 Tesla Scanning: MRI/MRS of glioma and non-glioma patients.
  Interventions: Device: 3 Tesla scanning

INTERVENTIONS:
Device: 3 Tesla scanning — Approximately 38 brain tumor patients with IDH mutated gliomas and 50 patients with non-glioma disease will be scanned.
  Other Names: 3T MRI/MRS

SUMMARY:
The Investigators will examine the disease specificity of 2-hydroxyglutarate in non-glioma brain lesions, and the clinical utility of 2-hydroxyglutarate, glycine and citrate in IDH mutated gliomas and IDH wild type gliomas.

DETAILED DESCRIPTION:
Malignant gliomas represent the majority of primary brain tumors in adults and are among the most intractable tumors. Cancers reprogram their metabolism to meet the needs of rapid cell growth. Alterations in metabolite abundance may serve as biomarkers of malignancy, and the capability to monitor the changes non-invasively would have significant clinical utility in cancer. Gliomas often contain a specific metabolic activity that is predictive of the genotype and has predictive value with respect to tumor stage and patient survival. A high fraction of gliomas contain mutations in the metabolic enzymes, isocitrate dehydrogenase (IDH) 1 and 2. These heterozygous mutations are confined to the active site of the enzyme and result in a neomorphic activity that causes the mutant enzyme to produce an "oncometabolite", 2-hydroxyglutarate (2HG). Non-invasive identification of this onco-metabolite by MRS is therefore a major breakthrough in cancer research. Beyond simple detection of 2HG, our preliminary data show that 2HG is a remarkably sensitive biomarker for monitoring tumor progression and response to treatment in IDH mutated gliomas. Glycine (Gly) is a biomarker of tumor malignancy, as indicated in prior studies. Our data also indicate that citrate (Cit) is elevated in gliomas.

Over the course of this preliminary study, there has been crucial need for 3D evaluation of these onco-metabolites within the tumor mass. The Investigators will examine the clinical utility of 2HG, Gly and Cit, in a large cohort of subjects using multi-slice 2D MRSI at 3T. The specific aims include, first, an in-vivo MRS study for the disease specificity of 2HG (Aim 1). The Investigators will examine clinically proven non-glioma lesions that mimic glioma in clinical MRI. To increase the clinical applicability of the result, the Investigators will select non-enhancing brain diseases, given that IDH mutation occurs largely in grade-2 and -3 gliomas, which are often non-enhancing. Second, the Investigators will examine the clinical utility of 2HG, Gly, Cit and other metabolites in patients with IDH mutated gliomas (Aim 2). Third, the Investigators will examine the clinical utility of Gly, Cit and other metabolites in patients with IDH wild type gliomas (Aim 3). In Aim 2 and 3, the patients will undergo MRSI scans at multiple time points, and the Investigators will monitor the metabolic changes with tumor progression and in response to treatment. The Investigators anticipate our study will provide significant value in many aspects of management of gliomas. 3D evaluation of the cancer biomarkers using MRSI will provide biological insights for making the diagnosis of gliomas, tracking of infiltrative cells during follow up, and determining response to treatment. Success of the 2HG specificity study in non-glioma neurological diseases will provide an experimental evidence for use of non-invasive 2HG imaging as a triaging tool in the workup of a new brain mass.

ELIGIBILITY:
Inclusion Criteria:

Patients with brain tumors (55 subjects):

* Age > 18 years
* Males and females
* All races and ethnicity
* Patients must meet at least one of the 3 following criteria regarding brain tumor diagnosis:

  * Histological diagnosis of a brain tumor
  * Pre-operative brain MR imaging suggestive of a brain tumor
  * Radiographic diagnosis of brain tumor in an inoperable location (e.g. brainstem)
* Pretreatment evaluation required for eligibility include a medical history, physical examination, and neurological exam within 30 days prior to study entry.
* Patient must be able to provide study-specific consent prior to study entry and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization.

Karnofsky performance status > 70%

Patients with non-tumor neurological disorders (50 subjects):

* Males and females
* All races and ethnicities
* Patients with clinically-proven encephalitis (infections, autoimmune and paraneoplastic), demyelinating lesions, vascular lesions (subacute arterial infarct, venous infarct, and vasculitis), hamartomatous lesions, and malformations of cortical development.

Exclusion Criteria:

* Age under 18*.
* Cardiac pacemaker.
* Intracranial clips, metal implants, or external clips within 50 cm from the head.
* Metal in eye.
* Pregnancy.
* Claustrophobia.
* Obesity or any other factors that provide difficulty with supine pose in the magnet.
* Patients who are unable to provide informed consent.
* Patients who are pregnant or nursing.
* Patients with severe kidney dysfunction or uncontrolled cardiac dysfunction.
* Patients who are claustrophobic or have other contraindication to MRI, such as implanted pacemaker device, vascular cips, surgical slips, prosthetic valves, pacemakers, otologic implants.
* Patients with uncontrolled psychiatric manifestations of their brain tumor.
* Children (age < 18) are excluded from the study plan because the incidence of astrocytomas and glioblastoma in children is far less than in adults. Although children frequently develop brain tumors, the glial tumors are most often pilocytic astrocytomas. In addition, enrollment of adults will be beneficial for the MRS sequence validation tests in healthy subjects since adults can remain motionless during the MR scans compared to children, giving minimal motion artifacts om the MR data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and over with brain tumors and patients 18 years of age and over with non-tumor neurological disorders.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of 2-hydroxygluterate (2HG) biomarker in 30 patients with clinically-proven brain metastasis, multiple sclerosis, epilepsy, stroke, or encephalitis using magnetic resonance spectroscopy (MRS). | 8 scans, average 36 months
  The investigators anticipate the study will provide significant value in many aspects of management of gliomas. 3D evaluation of the cancer biomarkers using MRSI will provide biological insights for making the diagnosis of gliomas, tracking of infiltrative cells during follow up, and determining response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Changho Choi, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No